CLINICAL TRIAL: NCT04601610
Title: An Open, Multi-center, Ib/II Clinical Trial of KN046 Combined With Ningatinib in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: KN046 Combined With Ningatinib in the Treatment of Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor's development strategy adjustment resolution is terminated
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN046-208
Record Dates: First submitted 2020-10-19; First posted 2020-10-26 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-05

CONDITIONS: Advanced HCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Subjects who have not received first-line system treatment previously;
  Interventions: Drug: KN046 （PD-L1/CTLA4 BsAb）; Drug: Ningetinib Tosylate（multi-target TKI）
- Cohort 2 (Experimental): Subjects who have received at least first-line system treatment
  Interventions: Drug: KN046 （PD-L1/CTLA4 BsAb）; Drug: Ningetinib Tosylate（multi-target TKI）

INTERVENTIONS:
Drug: KN046 （PD-L1/CTLA4 BsAb） — KN046 5mg/kg Q3W
Drug: Ningetinib Tosylate（multi-target TKI） — ningtinib QD, dose will be decided by investigator

SUMMARY:
This study is an open, multi-center clinical trial, the purpose is to study the safety and preliminary efficacy of KN046 combined with Ningatinib in subjects with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
The study consists of dose escalation and dose expansion, the mTPI-2 (Modified Toxicity Probability Interval) will be used for dose exploration. The preset dose of KN046 is 5 mg/kg Q3W and the preset dose of ningatinib is 10 mg (rapid titration), 20 mg QD, 30 mg QD, and 40 mg QD.Dose expansion will be divided into two cohorts, cohort 1 will enroll subjects who have not received system therapy and cohort 2 will enroll subjects who have previously received at least first-line system therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of hepatocellular carcinoma confirmed by histology or cytology；
* Barcelona Clinic Liver Cancer (BCLC) Stage B or C；
* ECOG performance status: 0-1；
* Child Pugh score≤7；
* Enough organ function；
* Has at least one measurable lesion based on RECIST 1.1；
* Life expectancy ≥3 months；
* Patients must be able to understand and willing to sign a written informed consent document；

Exclusion Criteria:

* Fibrous lamina hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma etc;
* Past or present hepatic encephalopathy; or Budd-Chiari syndrome; or Tumor thrombus invasion at the main portal vein (Vp4), inferior vena cava or heart involvement;
* Subjects who have previously received immune checkpoint inhibitors (such as anti-PD-1/L1, CTLA-4, etc.); or have a history of ≥ grade 3 immune-related adverse reactions; or hyperprogressive after immunotherapy previously；
* Subjects who have received liver local treatment (transcatheter chemoembolization, transcatheter embolization, hepatic artery perfusion, radiotherapy, radioembolization or ablation) within 4 weeks before administration;
* Subjects who need corticosteroids or immunosuppressive agents for systemic therapy;
* Any previous or current active autoimmune disease or history of autoimmune disease;
* History of liver transplantation;
* History of interstitial lung disease or non-infectious pneumonia;
* History of allergic reactions to related drugs;
* LVEF< 50% or LLN
* Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients undergoing total gastrectomy;
* With serious systemic diseases such as heart disease and cerebrovascular disease, and the condition is unstable or uncontrollable;
* Subjects with clinically significant gastrointestinal bleeding or thrombosis or embolic events within 6 months;
* Untreated hepatitis infection: HBV DNA>2000IU/ml or10000 copies/ml, HCV RNA> 1000copy/ml, both HbsAg and anti-HCV body are positive;
* Evidence of active pulmonary tuberculosis (TB);
* Positive test of immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
* Pleural effusion, ascites and pericardial effusion with clinical symptoms or needing drainage;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
DLT | 1 months
  Dose limit toxicity
ORR | 1 years
  objective response rate (ORR) based on the RECIST 1.1 by investigator

SECONDARY OUTCOMES:
PFS | 1.5 years
  progression free survival
OS | 3 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: JianMing Xu, Doctor, Principal Investigator — 301 Hospital of PLA，Beijing，China; ShanZhi Gu, Doctor, Principal Investigator — Hunan Cancer Hospital; YuXian Bai, Doctor, Principal Investigator — Harbin Medical University
Locations (1):
- Chinese Pla General Hospital Chinese Pla Medical School, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No